CLINICAL TRIAL: NCT06315868
Title: Breast Cancer Subtype Characterization Through Patient's Derived Organoids". (BCinsightPDO)
Brief Title: Breast Cancer Subtype Characterization Through Patient's Derived Organoids.
Acronym: BCinsightPDO
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5590
Record Dates: First submitted 2023-05-11; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer; Organoids
Keywords: breast cancer; new drugs; organoids
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Bioptic samples of Breast Cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Development of tools to predict patients chemo-sensitivity and identification of corresponding biomarkers is an urgent challenge for BC patients lacking targeted therapies, such as TNBC, or for patients experiencing relapse after adjuvant chemotherapy or targeted therapies.

The refinement of 3D-cultivation techniques, experienced in the last decade, has allowed cultivation of patients-derived cancer cells in organotypic structures, named patient-derived organoids (PDO), which preserve histologic, genomic and transcriptomic features of primary tumors. PDO allow propagation, pharmacological treatment and genetic manipulation of patients-derived cancer cells in a close to physiology setting, thus representing a promising tool in the development of personalized therapies

DETAILED DESCRIPTION:
PDO have been shown to efficiently recapitulate ex-vivo the in vivo response to hormonal treatment of BC patients. These observations point to PDO as potential valuable tools for a rapid, personalized prospective evaluation of patient-specific chemo-sensitivity. Moreover, PDO can represent a valuable ex-vivo platform for screening new treatments, or combination of current treatments, in a medium-to-high-throughput fashion. Thus, development of a stable collection of PDO representing the heterogeneity of BC subtypes, including the evolution of recurrent disease, represents an extremely useful resource for both prospective and retrospective studies aimed at understanding the molecular phenotype associated with chemoresistance.

ELIGIBILITY:
Inclusion Criteria:

* women diagnosed with primary BC, eligible for surgical resection of the tumor according to national and international guidelines.

age between 18 and 70 years; newly diagnosed breast neoplasms, tumor size of at least 1.5 cm diameter.

Exclusion Criteria:

breast cancer diagnosed during pregnancy, neoadiuvant chemotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible population includes women diagnosed with primary BC, eligible for surgical resection of the tumor according to national and international guidelines. Each case will be discussed, before surgery, at the multidisciplinary tumor board for BC of the Fondazione Policlinico A. Gemelli, IRCCS.
  All women will be required to sign written informed consent to enter the study. The study design has considered following inclusion criteria: age between 18 and 70 years; newly diagnosed breast neoplasms, tumor size of at least 1.5 cm diameter.
Sampling Method: Probability Sample
Enrollment: 306 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
evaluate the histological and molecular conformity (yes/no) between PDO and matched primary and/or recurrent BC sample, in order to develop a live biobank of ER/PR+, HER2+ and TNBC PDO. | 36 months
  Part of each surgical specimen will be used to obtain PDOs according to established procedures, part will be fixed and paraffin embedded for histological analysis and part will be flash-frozen for DNA, RNA and protein analyses. At first passages, organoids will be characterized for histologic and cytologic features. PDOs that faithfully recapitulate features of the matched primary tumor will be analysed for genomic features and splicing-sensitive transcriptomic signatures by next generation sequencing (NGS). Dichotomic variable: Yes (conform)/No (not conform)
evaluate the sensitivity of ER/PR+, HER2+ and TNBC PDO to novel therapeutic agents in clinical trials for BC or other cancer types | 42 months
  PDO will be tested for their susceptibility to the therapeutic agents administered to the corresponding patients and/or to novel therapeutic agents in clinical trials for BC or other cancer types by performing cell viability assays and clonogenic potential assay before and after treatments. Sensitivity to the tested drugs will be evaluated on the basis of the known maximal plasma concentration of the drug (Cmax): sensitive if survival is <50% at Cmax dose; resistant if survival is >50% at Cmax dose. Dichotomic variable: Yes (sensitive)/No (resistant)

SECONDARY OUTCOMES:
test the sensitivity of PDO to splicing-targeting treatments, either alone or in combination with other therapies | 42 months
  PDO derived from primary and recurrent BC patients will be evaluated for sensitivity to splicing-targeting drugs, administered either alone or in combination with standard chemotherapy. Sensitivity to the splicing-targeting drugs tested will be evaluated on the basis of the known EC50 of the drug for its molecular target: sensitive if survival is <50% at EC50 dose; resistant if survival is >50% at EC50 dose. Dichotomic variable: Yes (sensitive)/No (resistant). Combination index (CI) will be evaluated to assess synergic effects, with CI < 1 indicates synergism.
test the synergizing effects of agents splicing-targeting treatments to immunotherapies by co-culture experiments with autologous immune cells | 42 months
  PDO treated or not with the selected splicing inhibitor(s) will be exposed to PMBCs from the same patient previously stored under viable conditions, in presence or not of clinically available immune checkpoint inhibitors (anti-PD1 and anti-PD-L1 antibodies). Survival and proliferation assays will assess if treatment enhances the cytotoxic activity of PBMC towards cancer cells. Dichotomic variable: Yes/No

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Policlinico A. Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Harbeck N, Gnant M. Breast cancer. Lancet. 2017 Mar 18;389(10074):1134-1150. doi: 10.1016/S0140-6736(16)31891-8. Epub 2016 Nov 17. PMID 27865536
- [Background] Garrido-Castro AC, Lin NU, Polyak K. Insights into Molecular Classifications of Triple-Negative Breast Cancer: Improving Patient Selection for Treatment. Cancer Discov. 2019 Feb;9(2):176-198. doi: 10.1158/2159-8290.CD-18-1177. Epub 2019 Jan 24. PMID 30679171
- [Background] Denkert C, Liedtke C, Tutt A, von Minckwitz G. Molecular alterations in triple-negative breast cancer-the road to new treatment strategies. Lancet. 2017 Jun 17;389(10087):2430-2442. doi: 10.1016/S0140-6736(16)32454-0. Epub 2016 Dec 7. PMID 27939063
- [Background] Liedtke C, Mazouni C, Hess KR, Andre F, Tordai A, Mejia JA, Symmans WF, Gonzalez-Angulo AM, Hennessy B, Green M, Cristofanilli M, Hortobagyi GN, Pusztai L. Response to neoadjuvant therapy and long-term survival in patients with triple-negative breast cancer. J Clin Oncol. 2008 Mar 10;26(8):1275-81. doi: 10.1200/JCO.2007.14.4147. Epub 2008 Feb 4. PMID 18250347
- [Background] Kornblihtt AR, Schor IE, Allo M, Dujardin G, Petrillo E, Munoz MJ. Alternative splicing: a pivotal step between eukaryotic transcription and translation. Nat Rev Mol Cell Biol. 2013 Mar;14(3):153-65. doi: 10.1038/nrm3525. Epub 2013 Feb 6. PMID 23385723
- [Background] Pagliarini V, Naro C, Sette C. Splicing Regulation: A Molecular Device to Enhance Cancer Cell Adaptation. Biomed Res Int. 2015;2015:543067. doi: 10.1155/2015/543067. Epub 2015 Jul 26. PMID 26273627
- [Background] Chabot B, Shkreta L. Defective control of pre-messenger RNA splicing in human disease. J Cell Biol. 2016 Jan 4;212(1):13-27. doi: 10.1083/jcb.201510032. PMID 26728853
- [Background] Karni R, de Stanchina E, Lowe SW, Sinha R, Mu D, Krainer AR. The gene encoding the splicing factor SF2/ASF is a proto-oncogene. Nat Struct Mol Biol. 2007 Mar;14(3):185-93. doi: 10.1038/nsmb1209. Epub 2007 Feb 18. PMID 17310252
- [Background] Hsu TY, Simon LM, Neill NJ, Marcotte R, Sayad A, Bland CS, Echeverria GV, Sun T, Kurley SJ, Tyagi S, Karlin KL, Dominguez-Vidana R, Hartman JD, Renwick A, Scorsone K, Bernardi RJ, Skinner SO, Jain A, Orellana M, Lagisetti C, Golding I, Jung SY, Neilson JR, Zhang XH, Cooper TA, Webb TR, Neel BG, Shaw CA, Westbrook TF. The spliceosome is a therapeutic vulnerability in MYC-driven cancer. Nature. 2015 Sep 17;525(7569):384-8. doi: 10.1038/nature14985. Epub 2015 Sep 2. PMID 26331541
- [Background] Chan S, Sridhar P, Kirchner R, Lock YJ, Herbert Z, Buonamici S, Smith P, Lieberman J, Petrocca F. Basal-A Triple-Negative Breast Cancer Cells Selectively Rely on RNA Splicing for Survival. Mol Cancer Ther. 2017 Dec;16(12):2849-2861. doi: 10.1158/1535-7163.MCT-17-0461. Epub 2017 Sep 6. PMID 28878028
- [Background] Stricker TP, Brown CD, Bandlamudi C, McNerney M, Kittler R, Montoya V, Peterson A, Grossman R, White KP. Robust stratification of breast cancer subtypes using differential patterns of transcript isoform expression. PLoS Genet. 2017 Mar 6;13(3):e1006589. doi: 10.1371/journal.pgen.1006589. eCollection 2017 Mar. PMID 28263985
- [Background] Trincado JL, Sebestyen E, Pages A, Eyras E. The prognostic potential of alternative transcript isoforms across human tumors. Genome Med. 2016 Aug 17;8(1):85. doi: 10.1186/s13073-016-0339-3. PMID 27535130
- [Background] Kahles A, Lehmann KV, Toussaint NC, Huser M, Stark SG, Sachsenberg T, Stegle O, Kohlbacher O, Sander C; Cancer Genome Atlas Research Network; Ratsch G. Comprehensive Analysis of Alternative Splicing Across Tumors from 8,705 Patients. Cancer Cell. 2018 Aug 13;34(2):211-224.e6. doi: 10.1016/j.ccell.2018.07.001. Epub 2018 Aug 2. PMID 30078747